CLINICAL TRIAL: NCT02774616
Title: BIO|MASTER.Ilivia Family / Plexa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TA111
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure; Tachyarrhythmia
MeSH Terms: conditions — Heart Failure; Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ilivia ICD Family (Other): Implant of the new Ilivia ICD Family. Device measurements, pre-defined programming and Adverse Event Reporting
  Interventions: Device: Ilivia ICD Family
- Plexa ICD lead (Other): Implant of the new Plexa ICD lead. Device measurements and Adverse Event Reporting
  Interventions: Device: Plexa ICD lead
- Ilivia ICD and Plexa lead (Other): Implant of the new Ilivia ICD Family and the new Plexa lead. Device measurements, pre-defined programming and Adverse Event Reporting
  Interventions: Device: Ilivia ICD Family; Device: Plexa ICD lead

INTERVENTIONS:
Device: Ilivia ICD Family — pre-defined device programming, measurements and follow-up schedule
  Arms: Ilivia ICD Family; Ilivia ICD and Plexa lead
Device: Plexa ICD lead — predefined follow-up schedule
  Arms: Ilivia ICD and Plexa lead; Plexa ICD lead

SUMMARY:
Post-Market Clinical Follow-up of the new Ilivia ICD Family and the new Plexa right ventricular lead to fulfill requirements by the notified body and to support regulatory approval outside of the CE region

ELIGIBILITY:
Inclusion Criteria:

* Standard indication for ICD or CRT-D therapy according to clinical practice
* De novo implantation or upgrade/exchange (group A only) from existing ICD, CRT-D or pacemaker implant
* Patient is able to understand the nature of the clinical investigation and provides written informed consent
* Patient is able and willing to complete all routine study visits at the investigational site
* Patient accepts Home Monitoring concept
* Age ≥ 18 years

Exclusion Criteria:

* Contraindication to ICD or CRT-D therapy, respectively
* For CRT-D patients in group A only: physician not willing to activate MultiPole Pacing in the patient
* Cardiac surgical procedure planned within 6 months after implantation (including also interventional procedures like ablation, valve replacement etc.). Procedures to occur during or prior to implantation are not exclusionary.
* Expected to receive heart transplant or ventricular assist device within 6 months
* Life expectancy less than 6 months
* Participation in any other interventional clinical investigation
* Pregnant or breastfeeding at time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Sticherling, Prof. Dr., Study Chair — Universitätsspital Basel
Locations (25):
- Australia (2):
  - Liverpool Hospital, Liverpool
  - Nambour General Hospital, Nambour
- Universitätsklinikum St. Pölten, Sankt Pölten, Austria
- Odense University Hospital, Odense, Denmark
- CHU Brest, Brest, France
- Germany (10):
  - Hufeland Klinikum GmbH, Bad Langensalza
  - HDZ NRW Bad Oeynhausen, Bad Oeynhausen
  - Städtisches Klinikum Brandenburg GmbH, Brandenburg
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Westpfalz-Klinikum Kaiserslautern, Kaiserslautern
  - Hegau-Bodensee-Klinikum Singen, Singen
  - Universitätsklinikum Würzburg, Würzburg
- Israel (2):
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- National Heart Center Singapore, Singapore, Singapore
- Spain (3):
  - Hospital de Bellvitge, Barcelona
  - Hospital de Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de Macarena, Seville
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonspital Luzern, Lucerne

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 292 patients completed the informed consent process and signed the informed consent sheet.
Pre-assignment Details: 278 patients received one or more study devices implanted. 14 enrolled patients did not receive a study device and were excluded from the analysis. Reasons were implantation of other devices than the study devices (N = 8), no implantation of any device for different reasons (N = 5), or withdrawal of consent before implantation (N = 1).
Groups:
- Ilivia ICD and Plexa ICD Lead: Implant of the new Ilivia ICD and the new Plexa ICD lead
Period: Overall Study
Arm/Group | Ilivia ICD Family | Plexa ICD Lead | Ilivia ICD and Plexa ICD Lead
Started | 95 | 167 | 16
Died | 6 | 3 | 1
Withdrew Consent | 3 | 3 | 0
Lost to FU | 2 | 0 | 0
Device Explanted | 2 | 1 | 1
Other | 2 | 4 | 1
Completed | 80 | 156 | 13
Not Completed | 15 | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Ilivia ICD and Plexa ICD Lead: Implant of the new Ilivia ICD Family and the new Plexa ICD lead. Device measurements, pre-defined programming and Adverse Event Reporting
  Pre-defined device programming, measurements and follow-up schedule
- Total: Total of all reporting groups
Arm/Group | Ilivia ICD Family | Plexa ICD Lead | Ilivia ICD and Plexa ICD Lead | Total
Number analyzed (Participants) | 95 | 167 | 16 | 278
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [56 to 74] | 64 [57 to 72] | 71 [58 to 74.5] | 65 [57 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 29 | 5 | 51
  Male | 78 | 138 | 11 | 227
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Ilivia Family Related SADE-free Rate Through 3 Months
Description: This endpoint measures the percentage of patients without serious adverse device effect (SADE) related to the ICD device
Time Frame: 3 months
Population: These are all patients who either had a primary endpoint or who had reached 3 months of follow-up, or both.
Measure: Count of Participants; unit: Participants
Groups:
- Ilivia Arm; Ilivia ICD and Plexa ICD Lead: This endpoint was evaluated in patients of the Iliva arm and the Ilivia and Plexa arm combined
Arm/Group | Ilivia Arm | Ilivia ICD and Plexa ICD Lead
Number analyzed (Participants) | 92 | 12
Participants | 91 | 12
Statistical Analysis 1: Comparison: Ilivia Arm; Serious Adverse Device Effects (SADE) possibly or securely related to the Ilivia ICD family until the 3- month follow-up are counted for this primary endpoint. The following hypothesis has been defined: Ho: SADE-free rate through 3 months post-implant ≤ 90.0% Ha: SADE-free rate through 3 months post-implant > 90.0%; Test type: Non-Inferiority — A rejection of the null hypothesis (Ho) would demonstrate evidence that the complication-free rate is greater than 90.0% in the population; p = 0.0004, exact binomial

2. Primary Outcome: Plexa Related SADE-free Rate Through 6 Months
Description: This endpoint measures the percentage of patients without serious adverse device effect (SADE) related to the "Plexa" lead
Time Frame: 6 months
Population: These are all patients who either had an endpoint or who reached 6 months of follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Plexa Arm; Ilivia ICD and Plexa ICD Lead: This endpoint was evaluated in patients of the Plexa arm and of the Ilivia ICD and Plexa ICD lead arm combined
Arm/Group | Plexa Arm | Ilivia ICD and Plexa ICD Lead
Number analyzed (Participants) | 136 | 13
Participants | 133 | 12
Statistical Analysis 1: Comparison: Plexa Arm; Serious Adverse Device Effects (SADE) possibly or securely related to the Plexa ICD lead until the 6-month follow-up are counted for this primary endpoint. The following hypothesis has been defined: Ho: SADE-free rate through 3 months post-implant ≤ 90.0% Ha: SADE-free rate through 3 months post-implant > 90.0%; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0019, exact binomial

3. Secondary Outcome: Percentage of Patients With Successful Fast Ventricular Arrhythmia Conversion by ATP One-shot at 6-month Follow-up
Description: Of all patients with spontaneous ventricular arrhythmia detected in the VF zone, and treated by "ATP-one-shot", the percentage of patients with at least one successful termination will be determined
Time Frame: 6 months
Population: Only 5 patients had spontaneous ventricular arrhythmia detected in the VF zone.
Measure: Count of Participants; unit: Participants
Groups:
- Ilivia Arm: This endpoint was evaluated in patients of the Iliva arm with spontaneous ventricular arrhythmia detected in the VF zone
Arm/Group | Ilivia Arm
Number analyzed (Participants) | 5
Participants | 1

4. Secondary Outcome: Rate of Appropriate Right Ventricular Sensing at 3-month Follow-up
Description: The investigator is asked whether the sensing function of the Pleaxa lead in the right ventricle is appropriate
Time Frame: 3 months
Population: Patients in whom this endpoint was not evaluated did not attend the 3-months follow-up or the data were not recorded
Measure: Count of Participants; unit: Participants
Groups:
- Plexa Arm: This endpoint was evaluated in patients of the Plexa arm only
Arm/Group | Plexa Arm
Number analyzed (Participants) | 145
Participants | 145
Statistical Analysis 1: Comparison: Plexa Arm; Test type: Non-Inferiority — This endpoint evaluates the rate of appropriate right ventricular sensing of all patients in which a sensing measurement was performed. The following hypothesis has been defined: Ho: Rate of appropriate sensing through 3 months post-implant ≤ 93.0% Ha: Rate of appropriate sensing through 3 months post-implant > 93.0%; p < 0.0001, exact binomial — A rejection of the null hypothesis (Ho) would demonstrate evidence that the rate of appropriate sensing is greater than 93.0% in the population

5. Secondary Outcome: Rate of Appropriate Right Ventricular Pacing at the 3 Months Follow-up
Description: The investigator is asked whether the pacing function of the Pleaxa lead in the right ventricle is appropriate
Time Frame: 3 months
Population: Patients in whom this endpoint was not evaluated did not attend the 3-months follow-up or the data were not recorded
Measure: Count of Participants; unit: Participants
Arm/Group | Plexa Arm
Number analyzed (Participants) | 150
Participants | 150
Statistical Analysis 1: Comparison: Plexa Arm; This secondary hypothesis evaluates the rate of appropriate right ventricular pacing of all patients in which a pacing measurement was performed. The following hypothesis has been defined: Ho: Rate of appropriate pacing through 3 months post-implant ≤ 93.0% Ha: Rate of appropriate pacing through 3 months post-implant > 93.0%; Test type: Non-Inferiority — A rejection of the null hypothesis (Ho) would demonstrate evidence that the rate of appropriate pacing is greater than 93.0% in the population; p < 0.0001, exact binomial

ADVERSE EVENTS:
Time Frame: Patients of the Ilivia group were followed for 3 months. Patients of the Plexa group were followed for 6 months.
Arm/Group | Ilivia ICD Family | Plexa ICD Lead
All-Cause Mortality (participants affected / at risk) | 6/111 | 6/183
Serious Adverse Events (participants affected / at risk) | 48/111 | 56/183
Other Adverse Events (participants affected / at risk) | 52/111 | 49/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ilivia ICD Family (N=111) | Plexa ICD Lead (N=183)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 3 (3) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 6 (7) | 5 (5)
Atrial flutter (Cardiac disorders) | 2 (2) | 1 (2)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiogenic shock (Vascular disorders) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Coronary artery disorders (Cardiac disorders) | 1 (2) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
decompensated heart failure/ cardiac decompensation (Cardiac disorders) | 9 (11) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Device issue (General disorders) | 8 (8) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Eye disorders NEC (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal disorders NEC (Gastrointestinal disorders) | 3 (3) | 3 (3)
General disorders and administration site conditions NEC (General disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 3 (3) | 7 (11)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Inappropriate phrenic nerve stimulation (General disorders) | 2 (2) | 0 (0)
Infections and infestations NEC (Infections and infestations) | 2 (2) | 2 (2)
Injury, poisoning and procedural complications NEC (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Investigations NEC (Investigations) | 1 (1) | 1 (1)
Metabolism and nutrition disorders NEC (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder NEC (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Nervous system disorders NEC (Nervous system disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (2) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5)
Pneumonia (Infections and infestations) | 2 (3) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Psychiatric disorders NEC (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal and urinary disorders NEC (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4) | 4 (4)
Reproductive system and breast disorders NEC (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders NEC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Worsening Heart Failure (Cardiac disorders) | 0 (0) | 3 (3)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ilivia ICD Family (N=111) | Plexa ICD Lead (N=183)
Adverse drug reaction (General disorders) | 4 (4) | 7 (7)
Allergic reaction (Immune system disorders) | 4 (4) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
decompensated heart failure/ cardiac decompensation (Cardiac disorders) | 2 (3) | 1 (1)
Device issue (General disorders) | 8 (9) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Eye disorders NEC (Eye disorders) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders NEC (Gastrointestinal disorders) | 1 (2) | 1 (2)
General disorders and administration site conditions NEC (General disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (2)
Hematoma (Vascular disorders) | 1 (1) | 2 (2)
Hepatobiliary disorders NEC (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Inappropriate phrenic nerve stimulation (General disorders) | 12 (18) | 7 (12)
Infections and infestations NEC (Infections and infestations) | 0 (0) | 2 (2)
Intraoperative venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Investigations NEC (Investigations) | 0 (0) | 2 (2)
Metabolism and nutrition disorders NEC (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder NEC (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Nervous system disorders NEC (Nervous system disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders NEC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Skin and subcutaneous tissue disorders NEC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
Unevaluable event (General disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Vascular disorders NEC (Vascular disorders) | 0 (0) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 4 (4)
Worsening Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT02774616/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT02774616/SAP_001.pdf